CLINICAL TRIAL: NCT07074808
Title: HRV Guided Accelerated Diagnostic Protocol for Chest Pain Patients - Randomised Control Trial (HRV-ADP RCT)
Brief Title: RCT aiTriage Chest Pain Risk Stratification
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: CIRB 2022-2323
Record Dates: First submitted 2025-06-29; First posted 2025-07-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chest Pain; Emergencies
Keywords: Triage; emergency medicine; risk stratification; AI
MeSH Terms: conditions — Chest Pain; Emergencies

STUDY DESIGN:
Intervention Model Description: ADP vs Standard
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRV-ADP (Experimental): Using aiTriage risk score for stratification
  Interventions: Device: aiTriage risk score
- Standard Control (No Intervention): Standard control (no AI risk score)

INTERVENTIONS:
Device: aiTriage risk score — Risk score generated by AI App aiTriage for chest pain patients
  Arms: HRV-ADP

SUMMARY:
Chest pain is one of the most common reasons people visit the Emergency Department (ED). While most cases are not serious, a small number may lead to life-threatening heart problems, known as Major Adverse Cardiac Events (MACE). Emergency staff need to quickly identify these high-risk patients, but current methods often take time, involve lab tests, and strain already busy EDs.

In Singapore, for example, SGH sees over 120,000 ED patients a year. In the U.S., chest pain accounts for around 8-10 million ED visits annually, yet fewer than 10% are ultimately diagnosed with MACE. Still, over half of chest pain patients undergo extensive and costly testing, adding up to $10-13 billion each year. This over-testing is done to avoid missing a critical case, but it's inefficient and stressful for both staff and patients.

Traditional risk scoring tools like TIMI, GRACE, HEART, and EDACS require time and blood test results, delaying early intervention. Waiting times in EDs can be 1-2 hours, during which patient conditions may worsen unnoticed.

To address this, we've developed aiTriage, a portable device that uses AI to analyze heart rate variability, ECG readings, blood pressure, and oxygen levels. It provides a real-time risk score within 5 minutes, helping doctors decide which patients need urgent care. Unlike current methods, aiTriage works without waiting for lab tests and can ease the load on EDs.

No existing devices offer real-time MACE risk scoring like aiTriage. Our previous studies show that this system outperforms standard tools and could transform how chest pain is managed in emergency care, saving time, money, and lives.

DETAILED DESCRIPTION:
Primary Aim

* To compare the admission rate defined as number of patients admitted/ all patients presenting to ED with chest pain (Inpatient admission or Emergency Observation Ward admission) of HRV guided accelerated diagnostic protocol (HRV-ADP) to the current standard protocol.
* To evaluate the implementation of HRV-ADP and understand the potential factors affecting implementation success in routine practice using the REAIM/PRISM framework

Secondary Aim

* To determine 30-day MACE between groups for discharged patients.
* To determine ED length of stay from registration to admission decision between groups.
* To calculate predicted aiTriage HRV-ADP admission rate vs actual (control group).

Primary Hypothesis - There will be a 10-20% reduction in admission rate with HRV-ADP comparing to the Standard protocol currently in practice.

Secondary Hypothesis

- There is no increase in Major Adverse Cardiac Events (MACE) between groups for discharged patients.

ELIGIBILITY:
Inclusion Criteria:

* All ED patients (≥21 years old) with chest pain suspected of having ACS will be eligible for being included in this study.

Exclusion Criteria:

* Patients who are not in sinus rhythm
* Patients who do not have mental capacity.
* Patients with unstable vital signs, STEMI, obvious ACS, and non cardiac cases like rib fractures, pneumothorax.
* Patients lost to follow- up or transferred to other hospitals within the 30 day time frame.
* Patients with a high percentage of artefacts and ectopics exceeding 30% of ECG recordings will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1120 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Admission rate | Throughout in ED, an average of 3 days
  [number of patients admitted] divided by [all patients presenting to ED with chest pain]

SECONDARY OUTCOMES:
30-day MACE | 30 days starting from admission to ED
  Any major adverse cardiac events occurred in ED/hospital till discharged/death
Hospital Length of Stay | Within hospital stay, an average of 7 days
  From ED registration date/time to ward admission decision between groups
HRV-ADP Admission Rate | within hospital stay, an average of 7 days
  Admission rate (Intervention group vs Control Group)

CONTACTS AND LOCATIONS:
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mahler SA, Burke GL, Duncan PW, Case LD, Herrington DM, Riley RF, Wells BJ, Hiestand BC, Miller CD. HEART Pathway Accelerated Diagnostic Protocol Implementation: Prospective Pre-Post Interrupted Time Series Design and Methods. JMIR Res Protoc. 2016 Jan 22;5(1):e10. doi: 10.2196/resprot.4802. PMID 26800789
- [Background] Ong ME, Goh K, Fook-Chong S, Haaland B, Wai KL, Koh ZX, Shahidah N, Lin Z. Heart rate variability risk score for prediction of acute cardiac complications in ED patients with chest pain. Am J Emerg Med. 2013 Aug;31(8):1201-7. doi: 10.1016/j.ajem.2013.05.005. Epub 2013 Jun 10. PMID 23763936
- See also: aiTriage clinical trial in Singapore — https://www.duke-nus.edu.sg/newshub/our-stories/aitriage